CLINICAL TRIAL: NCT01454414
Title: Preventing Exposure to Ticks and Tick-borne Illness in Outdoor Workers
Brief Title: Tick-borne Illness and Clothing Study
Acronym: TICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-1027
Record Dates: First submitted 2011-10-10; First posted 2011-10-19 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2014-05

CONDITIONS: Tick Bites; Tick-borne Illness
MeSH Terms: conditions — Tick Bites

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Permethrin Impregnated Uniforms (Experimental): Uniforms (including pants, shorts, shirts, socks, and hats) treated with long-lasting permethrin.
  Interventions: Other: Permethrin Impregnated Uniforms
- Placebo (No Intervention): Uniforms sent to Insect Shield, washed and refolded (no permethrin applied).

INTERVENTIONS:
Other: Permethrin Impregnated Uniforms — Uniforms treated with permethrin according to proprietary process used by Insect Shield, Inc.
  Other Names: Insect Shield
  Arms: Permethrin Impregnated Uniforms

SUMMARY:
The high risk of acquiring tick-borne diseases by outdoor workers is well documented. Workers most at risk include, foresters, park rangers, land surveyors and other outdoor workers have frequent exposure to tick-infested habitats. Many North Carolina state employees with outdoor occupations report multiple tick bites each year, which indicates that existing tick preventive strategies may be ineffective. The principal goal of this study is to assess whether the use of long-lasting permethrin impregnated uniforms can reduce the number of tick bites sustained by North Carolina outdoor workers.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Employee of NC Division of Forest Resources, the NC Division of Parks and Recreation, NC Wildlife Resources Commission, or NC County and Local Parks and Recreation who work in Central and Eastern North Carolina
* An average of 10 or more hours of outdoor work per week during tick season
* Self-reported prior work-related tick bites

Exclusion Criteria:

* Pregnancy
* Non-English speaking
* Known allergy to insecticides

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Meshnick, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Gillings School of Global Public Health, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Vaughn MF, Funkhouser SW, Lin FC, Fine J, Juliano JJ, Apperson CS, Meshnick SR. Long-lasting permethrin impregnated uniforms: A randomized-controlled trial for tick bite prevention. Am J Prev Med. 2014 May;46(5):473-80. doi: 10.1016/j.amepre.2014.01.008. PMID 24745637

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Permethrin Impregnated Uniforms | Placebo
Started | 79 | 80
Baseline: Subjects That Sent Uniforms | 67 | 66
Completed | 66 | 64
Not Completed | 13 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Permethrin Impregnated Uniforms | Placebo | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (9.2) | 38.8 (9.3) | 39.0 (9.2)
Sex/Gender, Customized [Number; unit: participants] — One subject did not provide information on gender.
  participants
    Female | 14 | 11 | 25
    Male | 52 | 55 | 107
Race/Ethnicity, Customized [Number; unit: participants] — Sixteen subjects did not provide race or ethnicity information.
  participants
    White | 56 | 58 | 114
    Black | 2 | 0 | 2
    Other | 0 | 1 | 1
Education, categorical [Number; unit: participants] — Two subjects did not provide education information on the baseline questionnaire.
  participants
    High school or less | 5 | 10 | 15
    Some college | 20 | 14 | 34
    Bachelor or graduate degree | 40 | 42 | 82
Work division, categorical [Number; unit: participants] — One subject did not provide information on work division.
  participants
    NC Forest service | 21 | 27 | 48
    NC Division of Parks and Recreation | 31 | 25 | 56
    NC Wildlife Resources Commission | 9 | 10 | 19
    NC Local or County Parks and Recreation | 5 | 4 | 9
Years in current position, continuous [Mean (Standard Deviation); unit: years] | 7.9 (6.7) | 8.2 (6.8) | 8.0 (6.7)
Tick bites in previous year, continuous [Mean (Standard Deviation); unit: tick bites] | 19.3 (32.0) | 19.6 (39.3) | 19.4 (35.8)
Previous diagnosis with tick-borne illness [Number; unit: participants] — Self-reported diagnosis with a tick-borne illness prior to enrollment in the study.
  participants
    Lyme disease | 4 | 4 | 8
    Rocky Mountain spotted fever | 6 | 7 | 13
    Ehrlichiosis | 2 | 3 | 5
    Anaplasmosis | 0 | 0 | 0
    Babesiosis | 0 | 0 | 0
Use of tick bite prevention measures [Number; unit: participants]
  Long pants | 62 | 62 | 124
  Long sleeves | 48 | 52 | 100
  Hat | 43 | 38 | 81
  Tucked or taped pant legs | 5 | 7 | 12
  Repellent on skin | 22 | 22 | 44
  Repellent on clothing | 38 | 35 | 73
  Tick checks after working outdoors | 58 | 60 | 118
Use of self-applied permethrin on clothing [Number; unit: participants] | 30 | 34 | 64

OUTCOME MEASURES:

1. Primary Outcome: Work Related Tick Bites
Description: Tick bites are defined as ticks attached to or embedded in the skin
Time Frame: Weekly for two years
Measure: Number; unit: tick bites
Arm/Group | Permethrin Impregnated Uniforms | Placebo
Number analyzed (Participants) | 66 | 64
tick bites | 265 | 780
Statistical Analysis 1: Comparison: Permethrin Impregnated Uniforms vs Placebo; Protective effectiveness (1 - the incidence rate ratio) and 95% CIs for comparing reported tick bites between the treatment and control groups were calculated using a GEE model with a Poisson distribution and log link, and included terms for treatment, year of follow-up, and the interaction of treatment and year of follow-up, with an offset variable for log outdoor work hours; Test type: Superiority or Other; p = 0.004, Poisson regression; Protective effectiveness= 1 - rate ratio = 0.646, 95% CI 2-sided [0.288 to 0.824]

2. Secondary Outcome: Seroconversion Against a Tick-borne Illness
Description: We will define seroconversion as one in which there is a 4-fold change in Immunoglobulin G class antibody titer between sera at enrollment, sera obtained after one year and/or sera obtained at study's end or between acute and convalescent sera for participants developing an acute illness. The antigens that will be used in the serologic assays include Ehrlichia chaffeensis (which would also detect antibodies to E. ewingii and Anaplasma phagocytophilum) and Rickettsia rickettsii (which would also detect antibodies to other spotted fever group rickettsiae).
Time Frame: Upon enrollment, after the first year, and after the second year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Permethrin Impregnated Uniforms | Placebo
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/66
Other Adverse Events (participants affected / at risk) | 0/67 | 2/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Permethrin Impregnated Uniforms (N=67) | Placebo (N=66)
Tick-borne illness (serologically confirmed) (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No